CLINICAL TRIAL: NCT03154047
Title: A Phase 2b Open-label Extension Study to Evaluate the Long-term Safety and Efficacy of NEOD001 in Subjects With Light Chain (AL) Amyloidosis Who Were Previously Enrolled in Study NEOD001-201 (PRONTO)
Brief Title: Study in Subjects With Light Chain (AL) Amyloidosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: NEOD001 program terminated due to lack of clinical benefit
Sponsor: Prothena Biosciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEOD001-OLE251
Record Dates: First submitted 2017-04-28; First posted 2017-05-15 (Actual); Results first posted 2018-12-12 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: AL Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — birtamimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label (Experimental): Open Label Study Drug NEOD001
  Interventions: Drug: NEOD001

INTERVENTIONS:
Drug: NEOD001 — humanized monoclonal antibody

SUMMARY:
The objective of this study is to evaluate the long-term safety and efficacy of NEOD001 in subjects with AL amyloidosis who have completed Study NEOD001-201.

DETAILED DESCRIPTION:
Global, multicenter, Phase 2b, open-label extension study of subjects with AL amyloidosis who had a hematologic response to first-line treatment for their amyloidosis (e.g., chemotherapy, autologous stem cell transplant [ASCT]) and completed Study NEOD001-201. Subjects in this study may receive concomitant chemotherapy. Subject screening will occur during the 28 days prior to the first administration of study drug, which may overlap with the last visit in Study NEOD001-201. If all eligibility requirements are met, the subject will be enrolled and Screening assessments will be completed. Study visits will occur every 28 days based on scheduling from Month 1 Day 1. A ±5-day window is allowed for visits starting after Month 1. Subjects who discontinue study drug before the End of Study Visit (EOS) should have an Early Treatment Discontinuation Visit 30 (±5) days after their final administration of study drug. Each subject's study participation may be up to 38 months or until the study is terminated, whichever occurs first. The study consists of a Screening Phase (1 month), Treatment Phase (36 months), and EOS Visit (30 [±5] days after the last dose).

ELIGIBILITY:
Inclusion Criteria:

1. Completed the End of Study Visit in Study NEOD001-201
2. Adequate bone marrow reserve, hepatic and renal function, as demonstrated by:

   * Absolute neutrophil count (ANC) ≥1.0 × 109/L
   * Platelet count ≥75 × 109/L
   * Hemoglobin ≥9 g/dL
   * Total bilirubin ≤2 × upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) ≤3 × ULN
   * Alanine aminotransferase (ALT) ≤3 × ULN
   * Alkaline phosphatase (ALP) ≤5 × ULN (except for subjects with hepatomegaly and isozymes specific to liver, rather than bone)
   * Estimated glomerular filtration rate (eGFR) ≥25 mL/min/1.73 m2 as estimated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation, or measured GFR ≥25 mL/min/1.73 m2
3. Systolic blood pressure 80-180 mmHg
4. Women of childbearing potential must have a negative pregnancy test during Screening and must agree to use highly effective physician-approved contraception from Screening to 90 days following the last study drug administration
5. Male subjects must be surgically sterile or must agree to use highly effective physician-approved contraception from Screening to 90 days following the last study drug administration
6. Ability to understand and willingness to sign an informed consent form prior to initiation of any study procedures

Exclusion Criteria:

1. Any new medical contraindication or clinically significant abnormality on physical, neurological, laboratory, vital signs, or electrocardiographic (ECG) examination (e.g., atrial fibrillation; with the exception of subjects for whom the ventricular rate is controlled) that precludes continuation or initiation of treatment with NEOD001 or participation in the study
2. Symptomatic orthostatic hypotension that in the medical judgment of the Investigator would interfere with subject's ability to safely receive treatment or complete study assessments
3. Myocardial infarction, uncontrolled angina, uncontrolled ventricular arrhythmias, or ECG evidence of acute ischemia, within 6 months prior to the Month 1-Day 1 Visit
4. Severe valvular stenosis (e.g., aortic or mitral stenosis with a valve area <1.0 cm2) or severe congenital heart disease
5. ECG evidence of acute ischemia or active conduction system abnormalities with the exception of any of the following:

   * First degree atrioventricular (AV) block
   * Second degree AV block Type 1 (Mobitz Type 1/ Wenckebach type)
   * Right or left bundle branch block
   * Atrial fibrillation with a controlled ventricular rate (uncontrolled [i.e., >110 bpm] ventricular rate is not allowed [determined by an average of three beats in Lead II or 3 representative beats if Lead II is not representative of the overall ECG])
6. Has not recovered (i.e., equivalent to a Common Terminology Criteria for Adverse Events [CTCAE] ≥Grade 2) from the clinically significant toxic effects of prior anticancer therapy. Exception: subjects who have received treatment with a proteasome inhibitor such as bortezomib may have CTCAE Grade 2 neuropathy.
7. Received any of the following within the specified time frame prior to the Month 1-Day 1 Visit:

   * Oral or IV antibiotics, antifungals, or antivirals within 1 week, with the exception of prophylactic oral agents. Note: In the event that a subject requires the chronic use of antivirals, Medical Monitor permission is required for entry into the study.
   * Hematopoietic growth factors, transfusions of blood or blood products within 1 week
   * Chemotherapy, radiotherapy, HDAC inhibitors, or other plasma cell directed therapy within 2 weeks
   * ASCT within 4 weeks (i.e., ASCT is allowed if it occurred before enrollment in Study NEOD001-201 or after completion of Study NEOD001-201 if it was at least 4 weeks before Month 1-Day 1 of this study)
   * Major surgery within 4 weeks (or within 2 weeks following consultation with and approval of Medical Monitor)
   * Planned organ transplant during the study
   * Any investigational agent, other than NEOD001, within 4 weeks
   * Any experimental imaging agent directed at amyloid within 2 weeks
8. Active malignancy with the exception of any of the following:

   * Adequately treated basal cell carcinoma, squamous cell carcinoma, or in situ cervical cancer
   * Adequately treated Stage I cancer from which the subject is currently in remission and has been in remission for ≥2 years
   * Low-risk prostate cancer with Gleason score <7 and prostate-specific antigen <10 mg/mL
   * Any other cancer from which the subject has been disease-free for ≥2 years
9. History of Grade ≥3 infusion-related adverse events (AEs) or hypersensitivity to NEOD001
10. History of severe allergy to any of the components of NEOD001 such as histidine/L-Histidine, Trehalose, or Polysorbate 20
11. Currently known uncontrolled bacterial, viral, fungal, HIV, hepatitis B, or hepatitis C infection
12. Women who are breastfeeding
13. Any condition which could interfere with, or the treatment for which might interfere with, the conduct of the study or which would, in the opinion of the Investigator, unacceptably increase the subject's risk by participating in the study
14. Unable or unwilling to adhere to the study-specified procedures and restrictions
15. Subject is under legal custodianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (16):
  - City of Hope, Duarte, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mayo Clinic Hospital - Florida, Jacksonville, Florida
  - University of Chicago Medicine, Chicago, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic - Minnesota, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Westmead Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Eastern Health (Box Hill Hospital), Box Hill, Victoria
- Medizinische Universität Wien, Vienna, Austria
- France (2):
  - Hôpital Dupuytren - CHU Limoges, Limoges
  - Hôpital Pitié-Salpêtrière, Paris
- Germany (4):
  - Charité - Universitätsmedizin Berlin, Berlin
  - University of Duisburg-Essen, Essen
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
- Greece (2):
  - Alexandra General Hospital of Athens, Athens
  - University Hospital of Patras, Pátrai
- Hadassah Medical Center (HMC), Jerusalem, Israel
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
- Spain (2):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda
- United Kingdom (2):
  - Queen Elizabeth Hospital, Birmingham, England
  - The Royal Free Hospital, London, England

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- NEOD001 24 mg/kg: NEOD001, 24 mg/kg IV every 4 weeks for 36 months
Period: Overall Study
Arm/Group | NEOD001 24 mg/kg
Started | 80
Number of Patients Dosed | 80
Completed | 0
Not Completed | 80
Not completed — Death | 1
Not completed — Study terminated by sponsor | 76
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | NEOD001 24 mg/kg
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 2
  White | 74
  Other | 3
  Not Hispanic or Latino | 79
  Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: AEs are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome, or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Time Frame: Each subject's study participation may have been up to 36 months or until the study was terminated
Population: OLE Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- NEOD001 24 mg/kg: NEOD001, 24 mg/kg IV every 4 weeks
Arm/Group | NEOD001 24 mg/kg
Number analyzed (Participants) | 80
Participants
  Overall Number Baseline Subjects | 80
  Serious Adverse Events | 13
  Non-Serious Adverse Events | 57
  Death (all causes) | 1
  Death Resulting from Adverse Events | 1

ADVERSE EVENTS:
Time Frame: Initiation of study drug through study completion, up to 11 months
Description: AE that newly appears, increases in frequency, or worsens in severity following initiation of study drug and through the last study visit or up to 30 days after date of last dose, whichever is later.
Arm/Group | NEOD001 24 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/80
Serious Adverse Events (participants affected / at risk) | 13/80
Other Adverse Events (participants affected / at risk) | 28/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NEOD001 24 mg/kg (N=80)
Device related infection (Infections and infestations) | 1
Endocarditis bacterial (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic embolus (Infections and infestations) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NEOD001 24 mg/kg (N=80)
Upper respiratory tract infection (Infections and infestations) | 10
Fatigue (Gastrointestinal disorders) | 11
Oedema peripheral (General disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Nausea (Gastrointestinal disorders) | 7
Headache (Nervous system disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI, institution and the sponsor have agreed that the PI and institution may publish or disclose study results from their site after the earlier of (a) publication of the complete multicenter study results or (b) 18 months after database lock for the multicenter study. The sponsor has at least 45 days to review a proposed publication and may request deletion of confidential information and up to 60 days additional delay to obtain patent protection.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT03154047/SAP_000.pdf
  • Study Protocol (2017-01-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT03154047/Prot_001.pdf